CLINICAL TRIAL: NCT02704858
Title: An Open-Label, Phase 1/2A Dose Escalation Study of Safety and Efficacy of NEO100 in Recurrent or Progressive Grade III or Grade IV Gliomas With IDH1 Mutation
Brief Title: Safety and Efficacy Study in Recurrent or Progressive Grade III or IV IDH1 Mutated Glioma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neonc Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO100-01
Record Dates: First submitted 2016-01-27; First posted 2016-03-10 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma Multiforme
Keywords: recurrent glioblastoma; recurrent GBM
MeSH Terms: conditions — Glioblastoma | interventions — perillyl alcohol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NEO100 Phase 1 (Experimental): Intranasal delivery of NEO100 (perillyl alcohol) four times a day, escalation up to four different doses to determine maximum tolerated dose.
  Interventions: Drug: Perillyl alcohol
- NEO100 Phase 2A (Experimental): Intranasal delivery of NEO100 (perillyl alcohol) four times a day. Treatment of total of 25 patients at maximum tolerated dose.
  Interventions: Drug: Perillyl alcohol

INTERVENTIONS:
Drug: Perillyl alcohol — Intranasal administration
  Other Names: NEO100

SUMMARY:
This multi-site, Phase 1/2a clinical trial is an open-label study to identify the safety, pharmacokinetics, and efficacy of a repeated dose regimen of NEO100 (perillyl alcohol) for the treatment of patients with radiographically-confirmed progression of Grade IV glioma or recurrent primary or secondary Grade IV glioma. The study will have two phases, Phase 1 and Phase 2a. Phase 1 is a standard cohort dose escalation 3+3 design used to determine the maximum tolerated dose for Phase 2a. There will be up to 24 patients enrolled in Phase 1. There will be 25 patients enrolled in Phase 2a. For both phases of the study, NEO100 will be self-administered four times daily for a 28-day treatment cycles until disease progression, death or patient withdraw from study for any reason, whichever occurs first.

Version 10 of the protocol changed the inclusion criteria for Phase 2a to limit inclusion to those patients with progressive or recurrent primary or secondary Grade IV gliomas expressing IDH1 mutations. Prior to the protocol amendment, 4 patients were enrolled who were IDH1 wild-type. Therefore, an additional 28 patients will be recruited for a total of 32 patients enrolled into Phase 2a of this study to have 35 evaluable cases.

Version 12 of the protocol expanded the inclusion criteria for Phase 2a to include those patients with progressive or recurrent Grade III Astrocytoma expressing IDH1 mutations.

Review of the literature specific to these patients found the same expected time to progression and death. As a result, the number of patients to enroll remains 32 to have 35 evaluable cases.

DETAILED DESCRIPTION:
Malignant glioma, particularly glioblastoma multiforme (GBM, WHO grade IV astrocytic glioma) accounts for over half of all gliomas, which in turn account for 80% of all malignant brain and CNS tumors. In European and North American countries, the incidence rate is approximately four to five new cases per 100,000 people per year.

Most patients with glioblastoma are faced with a dismal prognosis. Advances in neurosurgery, radiation, and chemotherapy during the past decade have provided only small improvements in clinical outcome, with a 5-year survival rate remaining at less than 10%.The first-line treatment of GBM is usually surgery, both to confirm the diagnosis and to remove as much of the tumor as possible. Concurrent temozolomide with radiotherapy followed by adjuvant systemic temozolomide has produced a median survival of 14.6 to 16.6 months, and this regimen is now the standard of care for GBM, as well as grade III anaplastic glioma.

Regardless of the treatment regimen, the aggressive infiltration of glioblastoma throughout the brain typically produces progressive disability, ultimately leading to death in nearly all cases. Innovative treatment is urgently needed.

Molecular profiling is being used to separate patients with GBM into prognostic groups. A mutation affecting codon 132 of the isocitrate dehydrogenase 1 (IDH1) gene was found to occur in up to 12% of glioblastomas. A review of sequencing studies on large glioma patient cohorts have found IDH1 mutations present in 6% (range 3-16%).

IDH1 mutation is considered a definitive diagnostic molecular marker of glioblastomas and is considered more reliable and objective than clinical criteria. Long term outcome for patients with high-grade glioma including glioblastoma directly correlates to IDH1 mutation status. IDH1 mutated tumors have been associated with an improved outcome comparable to IDH1 wild-type tumors. IDH1 mutation has remained an independent favorable prognostic marker even after adjustment for age, grade, MGMT status, genomic profile and treatment in multivariate analysis. Median OS for glioblastoma patients following first recurrence is 9.8 months for IDH1 wildtype tumors versus 19.32 months for IDH1 mutated cancers. No increase in PFS was found.

Anaplastic astrocytoma is a rare, malignant brain tumor that arises from a subtype of glial cells that make up the majority of cells in the central nervous system, called astrocytes. Approximately 70-80% of WHO Grades II and III astrocytoma possess IDH mutations. In general, those diagnosed with initial grade III astrocytomas have a higher survival rate than patients with grade IV astrocytomas (5-year survival rate, Grade III, 71 participants, 49.2 ± 6.6 months vs. Grade IV, 216 patients, 9.6 ± 4.4 months). Interestingly, the presence of IDH mutations predict a favorable disease outcome with prolonged median survival in grade IV astrocytoma (IDH wild type: 15 months; IDH mutant: 31 months) and grade III anaplastic astrocytoma (IDH wild type: 20 months; IDH mutant: 65 months).

The reported median overall survival (OS) for glioblastomas is 14-15 months. Patients with initial diagnosis grade III astrocytoma have a considerably higher OS (45.2 ± 5.2 months with chemotherapy and radiotherapy, compared to 31.9 ± 2.7 months with no treatment), and progression free survival (PFS) (42.8 months treated with adjuvant temozolomide, compared to 19.0 months for people not treated with adjuvant temozolomide).

Patients with recurrent Grade III astrocytoma have effectively the same OS to grade IV tumors. A study carried out in 2018 showed 23 out of 100 patients experienced reoccurrence within an average time of 37 months after initial treatment and had an average OS after recurrence of 12.7 months. Additional research confirmed both that a high percentage of anaplastic astrocytomas reoccur and those that do occur have a median OS of approximately 10 months. Finally, 357 patients with highly anaplastic tumours were investigated between 1977 and 1989 (prior to the change in classification of brain tumors by the WHO). A total of 81 of these patients experienced tumour reoccurrence and required secondary treatment. The median OS for these patients was 53 weeks (13.2) months from the start of the secondary treatment. Based upon these studies, it is believed patients with IDH1 mutated recurrent or progressive Grade IV glioblastoma and IDH1 mutated recurrent or progressive Grade III astrocytoma have the same clinical prognosis with respect to progression free survival and overall survival and suitable for study in this protocol.

One reason for the poor prognosis of malignant glioma and astrocytoma patients is the difficulty of penetrating the blood brain barrier (BBB) with chemotherapy agents. Nasal brain delivery of chemotherapy offers a novel, paradigm shifting platform based on technology to deliver chemotherapy via inhalation to the brain tumor. The presumed mechanism of nasal brain delivery from preclinical rodent studies is thought to be via the olfactory and trigeminal nerves. Effective nasal brain delivery has been demonstrated in humans in other diseases. For example, Reger et al. have reported effective delivery of intranasal insulin for Alzheimer's disease.

NEO100 has been demonstrated to open the BBB in a reversible and nontoxic fashion in vitro and in vivo, enabling greatly increased brain entry of all tested therapeutics and was well tolerated in animals. Mechanistic studies revealed effects of NEO100 on different BBB transport pathways. An in vitro BBB, consisting of human astrocytes and brain endothelial cells, has been used to determine trastuzumab penetration when administered with NEO100, greatly increasing trastuzumab penetration. In vivo, IA NEO100-mediated BBB opening resulted in tumor-selective accumulation of trastuzumab , without detectable presence in normal brain tissue, along with increased presence of immune cell populations. IV delivery of trastuzumab or T-DM1 achieved significantly greater overall survival of tumor-bearing mice when combined with IA NEO100.

In a case lesson, after surgical removal of her recurrent GBM tumor, a patient received daily intranasal NEO100 therapy for more than 3 years before a second recurrence emerged. At that time, a final dose of NEO100 was given shortly before the tumor tissue was surgically removed, and the tissue was processed for high-performance liquid chromatography analysis of perillyl alcohol and its primary metabolite, perillic acid. Both molecules could readily be detected in the tumor tissue. This is the first demonstration of perillyl alcohol and perillic acid in brain tumor tissue from any patient. It reveals that intranasal administration of NEO100 is a valid approach to achieve delivery of this agent to a brain tumor. In view of the non-invasive and safe nature of this method, along with tentative indications of activity, these findings add confidence to the notion that intranasal administration of NEO100 holds potential as a new treatment option for brain-localized malignancies.

Perillyl alcohol, also called p-metha1,7-diene-6-ol,or 4-isopropenylcyclo-hexenecarbinol, is a monoterpene, isolated from the essential oils of lavender, peppermint, spearmint, and several other plants and synthesized by the mevalonate pathway. It has been previously demonstrated to have anti-cancer properties in preclinical studies in rodent models for a variety of cancers including mammary, pancreatic, and colon cancer. Although the exact mechanism of perillyl alcohol induced tumor regression is unknown, perillyl alcohol has been reported to modulate cellular processes that control cell growth and differentiation including G1 cell cycle arrest and induction of apoptosis.

Perillyl alcohol has also been shown to inhibit post-translational modification of proteins involved in signal transduction. It has been postulated that the anti-neoplastic activity of perillyl alcohol involves a decrease in the levels of isoprenylated Ras and Ras-related proteins, thereby reducing the physiological functioning of these proteins. Protein isoprenylation involves the post-translational modification of a protein by the covalent attachment of a lipophilic farnesyl isoprenoid group to a cysteine residue at or near the carboxyl terminus. Isoprenoid substrates for prenylprotein transferase enzymes include farnesyl pyrophosphate plus geranylgeranyl pyrophosphate, two intermediates in the mevalonate pathway. This action was attributed to the inhibition of farnesyl protein transferase activity. Farnesylation is the most critical part of the process that leads to the activation of Ras, and farnesyl transferase inhibitors exert their antitumor effect in part by inhibiting Ras-mediated signaling. A study revealed that H-Ras and K-Ras farnesylation were inhibited by perillyl alcohol.

Ras activity is elevated in malignant glioma tumors. Activated Ras stimulates other pathways essential for proliferation and progression through the cell cycle and inhibition of apoptosis in malignant gliomas. Moreover, the formation of malignant gliomas requires the cooperation of both Ras and Akt signaling. This cooperative effect has been demonstrated by somatic-cell gene transfer, during which transfer of either an activated form of K-Ras or Akt alone to neural progenitors was insufficient to form malignant glioma in vivo, but the combined effect of both pathways could initiate gliomagenesis. Thus, based on this known alteration in signal transduction involving K-Ras in malignant glioma, and its ability to induce cell cycle arrest and apoptosis, perillyl alcohol (NEO100) may be an attractive agent and warrants further clinical development.

Furthermore, intranasal delivery of NEO100 has the additional, potential benefit of direct drug delivery into the brain and avoiding systemic toxicity and first pass metabolism. It is believed the mechanism of action of NEO100 is similar in both patients with progressive or recurrent Grade IV gliomas who have IDH1 mutations and patients with progressive or recurrent Grade III astrocytomas who have IDH1 mutations making inclusion of both populations appropriate for this study.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in the study, a patient must meet all of the following inclusion criteria:

* Patient must have radiographically-confirmed progression of, or recurrent, primary or secondary Grade IV glioma, including infratentorial (brainstem, cerebellar) glioma (confirmed by biopsy) and subcortical glioma.
* Patient must have radiographically-confirmed progression of, recurrent, primary or secondary Grade III astrocytoma.
* All patients must be on a stable or decreasing dose of steroids for at least five days prior to the date of informed consent.
* Patient must have failed previous radiation treatment or combined treatment with temozolomide and radiation.
* If progression of disease occurs within 90 days of conformal radiation, the progression/recurrence must be outside of the radiation field or proven by biopsy/resection.
* Patient must be ≥ 18 years of age.
* Patient must have an ECOG performance status of 0-2 or KPS ≥ 60 (the latter for Phase 1 only).
* Patient must have an expected survival of at least three months.
* Patient must have a baseline MRI with gadolinium within 14 days of first administration of study drug.
* Patient must be willing to provide blood samples for pharmacokinetic study.
* If patient suffers from seizures, (s)he must be controlled on a stable dose of anti- epileptics for 14 days prior to the date of informed consent.
* Patient must have adequate organ and marrow function as defined below:
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SPGT)≤ 2.5 × institutional upper limit of normal
* Creatinine within normal institutional limits
* Female patients of child-bearing potential and male patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for 30 days prior to the first administration of study drug, for the duration of study participation, and for 90 days following completion of therapy. Should a female patient become pregnant, or suspect she is pregnant, while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* A negative serum pregnancy test will be required of all female patients of child-bearing potential within seven days prior to initiating study drug.
* A serum pregnancy test will be repeated immediately if pregnancy is suspected.
* Patient must have the ability to understand, and the willingness to sign, a written informed consent.

Phase 2a

In addition to meeting Inclusion Criteria for the Phase I portion of the study, patients eligible for participation in the Phase 2a portion of the study must additionally meet the following criteria:

• Patients must have a confirmed IDH1 mutation by reverse transcription polymerase chain reaction (rtPCR) or immunohistochemistry (unless continuing into the Phase 2a portion of the study from the Phase I portion of the study).

Exclusion Criteria

* If the patient meets any of the following criteria, the patient must not be enrolled:
* The size of the tumor is > 30mm (length x width), as assessed at the baseline (pre- study) MRI evaluation.
* The tumor is multi-focal, as assessed at the baseline (pre-study) MRI evaluation.
* Patient has completed chemo-radiation within the last 90 days prior to first administration of study drug, unless new contrast enhancement is outside of radiation field, or there is tissue proven recurrence or progression.
* Patient has had surgery within seven days prior to the date of informed consent.
* Patient has had any form of anti-cancer therapy or treatment within 28 days prior to first administration of study drug.
* Patient has not recovered from adverse events due to chemotherapy, immunotherapy, or radiation therapy administered more than 28 days prior to first administration of study drug.
* Patient has had prior treatment with bevacizumab, a chemotherapy wafer implant (Gliadel®), or any other FDA-approved anti-cancer therapy or treatment except temozolomide.
* Patient has had more than one recurrence or progression of his/her tumors.
* Patient has received any other investigational agents within 28 days prior to the first administration of study drug.
* Patient has had prior treatment with perillyl alcohol, administered either intravenously or intranasally.
* Patient has a history of allergic reactions attributed to perillyl alcohol.
* Patient has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Patient has a history of new diagnosis or treatment of cancer other than malignant glioma within five years prior to the date of informed consent, except for basal cell carcinoma or squamous cell carcinoma of the skin.
* Leptomeningeal involvement of the patient's tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Primary Outcome: Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Up to 6 months
Phase 2 Primary Outcome: Number of Participants Who Are Alive Each Month For 6 Months | Up to 6 months
Phase 2 Primary Outcome: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related To Treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chen, MD, PhD, Study Chair — NeOnc Technologies Holdings, Inc.; Josh Neman, PhD, Study Director — NeOnc Technologies Holdings, Inc.
Locations (11):
- United States (11):
  - University of Southern California, Los Angeles, California
  - Georgia Cancer Center (Augusta University), Augusta, Georgia
  - Ochsner Health, New Orleans, Louisiana
  - Atlantic Health (Overlook Medical Center), Summit, New Jersey
  - Northwell Health, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor Scott & White Health, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinic, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schonthal AH, Peereboom DM, Wagle N, Lai R, Mathew AJ, Hurth KM, Simmon VF, Howard SP, Taylor LP, Chow F, da Fonseca CO, Chen TC. Phase I trial of intranasal NEO100, highly purified perillyl alcohol, in adult patients with recurrent glioblastoma. Neurooncol Adv. 2021 Feb 12;3(1):vdab005. doi: 10.1093/noajnl/vdab005. eCollection 2021 Jan-Dec. PMID 33604574